CLINICAL TRIAL: NCT07142746
Title: Comparative Evaluation of Proximal Contact Tightness in Zirconia Crowns: Direct Digital Intraoral Scanning vs. Conventional Impressions Fabrication Method, A Randomized Control Trial.
Brief Title: Proximal Contact Tightness of Zirconia Crowns: Digital Intraoral Scanning vs Conventional Impressions
Acronym: PCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Seema Khattak, REGISTRAR PROSTHODONTICS, Armed Forces Institute of Dentistry, Pakistan
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Proximal Contact Tightness
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Proximal Contacts; Zirconia Crowns

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional impression (Active Comparator): One group will be receiving the impression for zirconia crowns by trays and conventional impression material.
  Interventions: Procedure: Conventional impression
- Digital Intra Oral Scanning (Experimental): One group will recieve digital intra oral scan for obtaining digital scan of anatomy of prepared teeth.
  Interventions: Procedure: Digital intra oral scanning

INTERVENTIONS:
Procedure: Digital intra oral scanning — One groups prepared teeth will be scanned by a digital intra oral scanner.
  Arms: Digital Intra Oral Scanning
Procedure: Conventional impression — One group will recieve impressions conventionally in a tray with dental impression polyvinly siloxane.
  Arms: Conventional impression

SUMMARY:
We will be comparing the proximal contacts of zirconia crowns and adjacent natural teeth in two groups. One receiving crowns fabricated via digital intra oral scanning means. And the other group recieving crowns fabricated via the dental impression method using trays and impression material.

DETAILED DESCRIPTION:
Subjects will be randomly assigned in two groups using a computer generated randomization list. Allocated subjects in groups will be concealed in an envelope. All clinical procedures of crown preparation and cementation will be performed by a single clinician with standard crown preparation guidelines to minimize variability. After standardized tooth preparation for full coverage ceramic crowns, one group will receive conventional impressions using polyvinyl siloxane (PVS) material in trays and other group will be scanned using intra oral digital scanner. Crowns for both groups will be fabricated in the same dental laboratory under standardized conditions.

Proximal and occlusal adjustments will be performed in the oral cavity before cementation at try in and crowns will be cemented using the same luting agent, GIC. After cementation proximal contact tightness will be assessed for the crowns by the digital force gauge at mesial and distal contacts and recorded for data compilation. The 0.05mm metal strip is inserted between the prosthesis and the adjacent natural tooth. The frictional force generated while removing the metal strip slowly in the buccal direction will be recorded on the screen of the customized digital force gauge. The frictional force generated will be considered equal to the proximal contact tightness and will be recorded in Newton (N). Proximal contact tightness will be recorded immediately after the crowns were cemented and at a recall after 10 days. These proximal contact tightness will be compared to see if there lies a significant difference in between the crowns fabricated from both impression techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking definitive full coverage ceramic crowns for molars.
* Patients in age group of 18- 47 years.
* Patients with healthy adjacent and opposing teeth.
* Patients with healthy periodontium.

Exclusion Criteria:

* Patients with grade 1 mobility in adjacent or opposing teeth.
* Patients with diastema in posterior teeth.
* Patients having severe malocclusion associated with traumatic occlusion.
* Patients with temporomandibular joint disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proximal contact tightness in terms of frictional force generated as shown on digital dynamometre in newtons at cementation day 1. | Day 1 at cementation of crown.
  Proximal contact tightness will be assesed when shimstock will be pulled out by a hook attached to a digital dynamometre. The frictional force generated in newtons will be assesed and noted at the day 1 of cementation.

SECONDARY OUTCOMES:
Proximal contact tightness of zirconia crowns in terms of frictional force in newtons as shown on digital dynamometre at the day 10. | At 10 days after receiving the treatment crown
  We will assess the proximal contact tightness of zirconia crowns with adjacent teeth as we pull shimstock with a hook attached to digital dynamometre and asses the frictional force generated in Newtons at the day 10 of cementation of crown.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Aleeha Zahoor Registrar Prosthodontics, Principal Investigator — Armed Forces Institute of Rawalpindi
Locations (1):
- Afid Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No